CLINICAL TRIAL: NCT05559580
Title: A Phase II, Randomised, Placebo-controlled, Double-blind, Parallel Group, Efficacy and Safety Study of at Least 48 Weeks of Oral BI 685509 Treatment in Adults With Progressive Systemic Sclerosis
Brief Title: A Study in People With Systemic Sclerosis to Test Whether Avenciguat (BI 685509) Has an Effect on Lung Function and Other Systemic Sclerosis Symptoms
Acronym: VITALISScE™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1366-0031; 2022-500332-11-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, investigators, central reviewers, and everyone involved in trial conduct or analysis or with any other interest in this double-blind trial will remain blinded regarding the randomised treatment assignments until the database is declared ready for analysis according to the sponsor's Standard Operating Procedures (SOPs).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Avenciguat (BI 685509) (Experimental): Avenciguat (BI 685509)
  Interventions: Drug: Avenciguat (BI 685509)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avenciguat (BI 685509) — Avenciguat (BI 685509)
  Arms: Avenciguat (BI 685509)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is open to adults aged 18 and older or above legal age who have systemic sclerosis. People can participate if they have a specific subtype called diffuse cutaneous systemic sclerosis. People with another subtype called limited cutaneous systemic sclerosis can also participate if they are anti Scl-70 antibody positive. Systemic sclerosis is also called scleroderma.

The purpose of this study is to find out whether a medicine called Avenciguat (BI 685509) helps people with scleroderma who have symptoms due to lung fibrosis or vascular problems.

Participants are put into 2 groups by chance. One group takes Avenciguat (BI 685509) tablets 3 times a day and the other group takes placebo tablets 3 times a day. Placebo tablets look like BI 685509 tablets but do not contain any medicine. Participants take the tablets for at least 11 months. Afterwards, participants can continue to take the tablets until the last participant has completed the 11-months treatment period. This means that the time in the study and duration of treatment is different for each participant, depending on when they start the study. At the beginning of the study, participants visit the study site every 2 weeks. The time between the visits to the study site gets longer over the course of the study. After the 11-months treatment period, participants visit the study site every 3 months.

During the study, participants regularly do lung function tests. The results are compared between the 2 groups to see whether the treatment works. The participants also regularly fill in questionnaires about their scleroderma symptoms. The doctors regularly check participants' skin condition and general health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent in accordance with International Council on Harmonisation (ICH) - Good Clinical Practice (GCP) and local legislation prior to admission to the trial.
2. Male or female patients aged ≥18 years at time of consent (or above legal age, e.g. United Kingdom (UK) ≥16 years).
3. Patients must fulfill the 2013 American College of Rheumatology/European Alliance of Associations for Rheumatology (ACR/EULAR) classification criteria for Systemic sclerosis (SSc).
4. Patients must be diagnosed with limited or with diffuse cutaneous SSc as defined by LeRoy et al. (R17 0149). Patients diagnosed with limited cutaneous SSc may be included if they are anti Scl-70 antibody positive.
5. Diffuse cutaneous SSc disease onset (defined by first non-RP symptom) in patients with diffuse cutaneous SSc must be within 7 years of Visit 1. Limited cutaneous SSc onset must be within 2 years of Visit 1.
6. Evidence of active disease, defined as having at least one of the following:

   * New onset of SSc within the last 2 years of Visit 1 OR
   * New skin involvement or worsening of two new body areas within 6 months of Visit 1 (out of the possible 17 body areas defined by Modified Rodnan Skin Score (mRSS) assessment, documented in clinical files) OR
   * New involvement or worsening of one new body area if either chest or abdomen within 6 months of Visit 1 OR
   * Worsening of skin thickening (e.g. ≥2 mRSS points) within 6 months of Visit 1 OR
   * ≥1 tendon friction rub
7. Elevated biomarkers on Visit 1 (screening) defined as at least one of the following:

   * C-reactive protein (CRP) ≥6 mg/L (≥0.6 mg/dL), OR
   * Erythrocyte sedimentation rate (ESR) ≥28 mm/h, OR
   * Krebs von den Lungen 6 (KL-6) ≥1000 U/mL If none of the three criteria are met or respective test results should not be available, the patient can be entered if the modified Disease Activity Index (mDAI) is ≥ 2.5.
8. Evidence of significant vasculopathy, defined as:

   * Active Digital ulcer (DU(s)) on Visit 1 OR
   * Documented history of DU(s), OR
   * Previous treatment of RP with prostacyclin analogues or ≥ 1 other medications, including calcium channel blockers, nitrates,, NO donors in any form, including topical; phosphodiesterase 5 (PDE5) inhibitors (e.g. sildenafil, tadalafil, vardenafil); nonspecific PDE5 inhibitors (theophylline, dipyridamole) OR
   * RP with elevated CRP ≥6 mg/L
   * If none of the four criteria above are met, the patient can be entered if the diagnosis of Interstitial lung disease (ILD) has been confirmed Further inclusion criteria apply.

Exclusion Criteria:

1. Any known form of pulmonary hypertension.
2. Pulmonary disease with FVC <50% of predicted. at screening.
3. Other autoimmune connective tissue diseases, except for fibromyalgia, scleroderma-associated myopathy and secondary Sjogren syndrome.
4. Diffusing capacity for carbon monoxide (DLCO) (haemoglobin corrected) <40% of predicted at screening.
5. Any history of scleroderma renal crisis within the last 6 months.
6. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (Chronic Kidney Disease Epidemiology (CKD-EPI) formula) or on dialysis at screening.
7. Cirrhosis of any Child-Pugh class (A, B or C).
8. Cholestasis at present, or Alkaline phosphatase (ALP) > 4 x Upper limit of normal (ULN), or ALP > 2 x ULN and Gamma-glutamyl transferase (GGT) > 3 x ULN at Screening.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of decline in forced vital capacity (FVC) (mL) over 48 weeks | 48 weeks.

SECONDARY OUTCOMES:
Absolute change from baseline in Modified Rodnan Skin Score (mRSS) at Week 48 in study participants with diffuse cutaneous systemic sclerosis (dcSSc) | At baseline and at week 48.
  To measure mRSS, skin thickness of the patient is rated by palpation using a scale of 0-3, with 0 = normal skin; 1= mild thickness; 2= moderate thickness and 3=severe thickness with an inability to pinch the skin into a fold (worst outcome).
Proportion of responders in study participants with diffuse cutaneous systemic sclerosis (dcSSc) based on the revised Composite Response Index in Systemic Sclerosis (CRISS) at Week 48 | At baseline and at week 48.
  Revised Composite Response Index in Systemic Sclerosis (CRISS) at Week 48 (Achievement of ≥ 20% improvement from baseline to week 48 in at least 3 of the 5 core set measures, except ≥ 5% in Forced Vital Capacity (FVC) percent predicted). The CRISS is a two-step composite index which includes in Step 2 the mRSS, FVC percent predicted, HAQ-DI, patient's global assessment and clinicians's global assessment. Step 1 in the ACR-CRISS version consists of the absence of significant worsening of interstitial lung disease, a new scleroderma renal crisis, left ventricular failure or pulmonary arterial hypertension. The revised version proposes that the absence of significant gastrointestinal dysmotility requiring parenteral or enteral nutrition and significant digital ischaemia requiring hospitalisation, gangrene or amputation are added to Step 1. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A higher score indicates greater improvement.
Absolute change from baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) score at Week 48 | At baseline and at week 48.
  HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area.
American College of Rheumatology Composite Response Index in Systemic Sclerosis (ACR-CRISS) score in study participants with diffuse cutaneous systemic sclerosis (dcSSc) at Week 48 | At week 48.
  The CRISS is a two-step composite index which includes in Step 2 the Modified Rodnan Skin Score (mRSS), FVC percent predicted, Health Assessment Questionnaire - Disability Index (HAQ-DI), patient's global assessment and clinicians's global assessment. Step 1 in the ACR-CRISS version consists of the absence of significant worsening of interstitial lung disease, a new scleroderma renal crisis, left ventricular failure or pulmonary arterial hypertension. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A higher score indicates greater improvement.
Absolute change from baseline in forced vital capacity (FVC) (mL) at Week 48 | At week 48.
Absolute change from baseline in forced vital capacity (FVC) (% predicted) at Week 48 | At baseline and at week 48.
Absolute change from baseline in the Patient Global Assesment (PGA) Visual Analog Scale (VAS) score at Week 48 | At baseline and at week 48.
  The PGA is a self-assessment on the patient's overall health in the prior 1 week using a 0-10 ordinal scale, with a higher score indicating a worse outcome.
Absolute change from baseline in the Clinician Global Assessment (CGA) Visual Analog Scale (VAS) score at Week 48 | At baseline and at week 48.
  Clinician assessment (CGA) on the patient's overall health in the prior 1 week using a 0-10 ordinal scale, with a higher score indicating a worst outcome.
Composite measure of Raynaud's phenomenon (RP) activity at Week 48 | Week 48.
Absolute change from baseline in Digital ulcer (DU) net burden at Week 48 | At baseline and at week 48.
Time to treatment failure | 48 weeks.
  Time to treatment failure, defined as the time to one of the following events (whichever occurs first) occurring over the 48-week and extended treatment period:
  * death,
  * absolute decline in percent-predicted forced vital capacity (FVC) ≥10% relative to baseline,
  * ≥25% increase in Modified Rodnan Skin Score (mRSS) and an increase in mRSS of >5 points,
  * initiation or dose change of immunomodulating/immunosuppressive therapy for clinically significant deterioration of Diffuse cutaneous systemic sclerosis (dcSSc)
Time to Modified Rodnan Skin Score (mRSS) progression (≥25% increase in mRSS and an increase in mRSS of >5 points) in study participants with diffuse cutaneous systemic sclerosis (dcSSc) | 48 weeks.
Proportion of study participants with diffuse cutaneous systemic sclerosis (dcSSc) with Modified Rodnan Skin Score (mRSS) progression (25% increase in mRSS and an increase in mRSS of >5 points) | 48 weeks.

CONTACTS AND LOCATIONS:
Locations (167):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Medvin Clinical Research-Covina-67001, Covina, California
  - Southern California Scleroderma and Rheumatology Center, Inglewood, California
  - University of California Los Angeles, Los Angeles, California
  - Medvin Clinical Research-Whittier-69033, Whittier, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Iris Research and Development, Plantation, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Argentina (7):
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - Hospital Britanico de Buenos Aires, CABA
  - STAT Research, CABA
  - Instituto de Investigación Clínica TyT, CABA
  - Psoriahue Medicina Interdisciplinaria S.R.L, CABA
  - Hospital Italiano de La Plata, La Plata
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- Austria (2):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - Ordensklinikum Linz GmbH, Linz
- Belgium (4):
  - ULB Hopital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Brazil (4):
  - SAPIENS - Instituto de Estudos e Pesquisa Clínica, Curitiba
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Hospital do RIM - UNIFESP, São Paulo
- Canada (4):
  - St. Paul's Hospital (Vancouver), Vancouver, British Columbia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Mount Sinai Hospital-Toronto-18157, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- Chile (2):
  - Centro Internacional de Estudios Clínicos (CIEC), Comuna de Recoleta
  - Clínica Dermacross S.A., Vitacura
- China (16):
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Affiliated Hospital Of Bengbu Medical College, Bengbu
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - The third affiliated hospital of Sun Yat-Sen University, Guangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Huashan Hospital, Fudan University, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital Affiliated Tongji Medical College Huazhong University of S & T, Wuhan
- Czechia (2):
  - Institute of Rheumathology Prague, Prague
  - Medical Plus s.r.o., Rheumatology Outpatient Clinic, Uherské Hradiště
- Aarhus University Hospital, Aarhus N, Denmark
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - TYKS, Turku
- France (7):
  - HOP Annecy-Genevois, Epagny Metz-Tessy
  - HOP Hôtel-Dieu, Nantes
  - Hôpital Cochin, Paris
  - HOP Pontchaillou, Rennes
  - HOP Civil, Strasbourg
  - Hôpital Rangueil - CHU de Toulouse, Toulouse
  - HOP Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum der Universität München AÖR, München
  - Westfälische Wilhelms-Universität Münster, Münster
- General Hospital of Athens "Laiko", Athens, Greece
- India (9):
  - St John's Medical College, Bangalore
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Sree Sudheendra Medical Mission, Kochi
  - Post Graduate Institute of Medical Education and Research, Kolkata
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institute, Maharashtra
  - Chopda Medicare and Research Centre Pvt Ltd, Maharashtra
  - All India Institute of Medical Sciences, New Delhi
  - Grant Medical Foundation, Ruby Hall Clinic, Pune
  - Krishna Institute of Medical Sciences, Secunderabad
- Israel (5):
  - Rambam Medical Center, Haifa
  - Bnai Zion Medical Center, Haifa, Haifa
  - Meir Medical Center, Kfar Saba
  - Western Galilee Hospital, Nahariya
  - The Chaim Sheba Medical Center Tel HaShomer, Ramat Gan
- Italy (10):
  - Ospedali Riuniti di Ancona, Ancona
  - A.O. Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera San Martino, Genova
  - Istituto Ortopedico G.Pini, Milan
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Fondazione Policlinico Universitario Campus Bio-medico, Roma
  - AOU Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Japan (8):
  - Japan Community Healthcare Organization Chukyo Hospital, Aichi, Nagoya
  - Hospital of the University of Occupational and Environmental Health, Fukuoka, Kitakyushu
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Kanazawa University Hospital, Ishikawa, Kanazawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - The University of Osaka Hospital, Osaka, Suita
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Malaysia (2):
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Selayang, Kuala Selangor
- Mexico (4):
  - Investigacion y Biomedicina de Chihuahua S.C., Chihuahua City
  - Centro Integral en Reumatologia, SA. de CV., Guadalajara
  - Medical Care & Research SA de CV, Mérida
  - Oaxaca Site Management Organization, S.C., Oaxaca City
- Netherlands (2):
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen
- Waikato Hospital, Hamilton, New Zealand
- Oslo Universitetssykehus HF, Rikshospitalet, Oslo, Norway
- Philippines (2):
  - Manila Doctors Hospital, Manila
  - St. Luke's Medical Center-Quezon-59457, Quezon City
- Poland (5):
  - Malopolska Clinical Research, Krakow
  - Medical Center Hetmanska, Poznan
  - National Medical Institute MSWiA, Warsaw
  - Prof Eleonora Reicher Memorial Institute of Rheumatology, Warsaw
  - Military Medical Institute- National Research Institute, Warsaw
- ULS de Almada -Seixal, E. P. E. - Hospital Garcia de Orta, Almada, Portugal
- Romania (8):
  - Bacau County Hospital, Bacau
  - C.M.D.T.A. NEOMED, Brasov, Brasov
  - Dr. Ion Cantacuzino Clinical Hospital, Bucharest
  - S.C. Policlinica CCBR S.R.L., Bucharest
  - St. Mary's Clinical Hospital, Bucharest
  - Cluj Napoca Clinical County Hospital, Cluj-Napoca
  - Aqua Clinic (AquaMed Consulting SRL- juridic), Constanța
  - SC Medaudio Optica SRL, Râmnicu Vâlcea
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - Hanyang University Medical Center, Seoul
- Spain (6):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Dr. Peset, Valencia
- Clinical Rheumatology Research Center Sahlgrenska, Gothenburg, Sweden
- Switzerland (2):
  - Kantonsspital St.Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Thailand (4):
  - Maharaj Nakom Chiangmai Hospital, Chiang Mai
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Muang
  - Ramathibodi Hospital, Ratchathewi
- Turkey (Türkiye) (2):
  - Akdeniz Universitesi Tip Fakultesi -ANTALYA-33606, Antalya
  - Firat University Hospital, Elâzığ
- United Kingdom (4):
  - Chapel Allerton Hospital, Leeds
  - Aintree University Hospital, Liverpool
  - Royal Free Hospital, London
  - Salford Royal, Salford

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Kaufman J, Nabozny G, Tran-Manh C, Liebel C, Zhou X, Daley LA, Wang CT, Ebenezer DL, Delic D, Wohnhaas CT, Trinh-Minh T, Distler JHW. Avenciguat: a novel soluble guanylate cyclase activator that affects multiple cell types to inhibit IFN-1 signalling and fibrosis. Rheumatology (Oxford). 2025 Aug 1;64(8):4738-4743. doi: 10.1093/rheumatology/keaf109. PMID 39985455
- [Derived] Khanna D, de Vries-Bouwstra J, Hoffmann-Vold AM, Kuwana M, Low AHL, Proudman S, Flack M, Kukreja A, Fagan N, Distler O. A Phase II study of avenciguat, a novel soluble guanylate cyclase activator, in patients with systemic sclerosis: Study design and rationale of the VITALISScE study. J Scleroderma Relat Disord. 2024 Nov 7;10(1):27-35. doi: 10.1177/23971983241291923. eCollection 2025 Feb. PMID 39544899
- See also: Related Info — http://www.mystudywindow.com